CLINICAL TRIAL: NCT02252185
Title: A Prospective, Multicenter, Randomized, Open-label, Controlled Study to Evaluate the Safety and Efficacy of a Spine Fusion System in Vertebral Body Fusion Surgery
Brief Title: A Clinical Study of a Spine Fusion System in Vertebral Body Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Medical (Suzhou) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPS-201303
Record Dates: First submitted 2014-09-24; First posted 2014-09-30 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-03

CONDITIONS: Disc Degenerative Disease; Spondylolisthesis; Spinal Fracture; Spinal Deformity; Spinal Stenosis; Spinal Tumor
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spinal Fractures; Spinal Stenosis; Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- China made spine fusion system (Experimental): patents in this arm will be implanted with Johnson&Johnson Medical Suzhou made Spine Fusion System.
  Interventions: Device: Johnson&Johnson Medical Suzhou made Spine Fusion System
- Imported spine fusion system (Active Comparator): patents in this arm will be implanted with Imported EXPEDIUM screws and OPAL cage .
  Interventions: Device: Imported EXPEDIUM screws and OPAL cage

INTERVENTIONS:
Device: Johnson&Johnson Medical Suzhou made Spine Fusion System — interventional device is Spine Fusion System that is manufactured by Johnson & Johnson Medical Suzhou Ltd.
  Arms: China made spine fusion system
Device: Imported EXPEDIUM screws and OPAL cage — Comparator in this study is active comparator.
  Arms: Imported spine fusion system

SUMMARY:
The primary objective of this study is to demonstrate that the efficacy and safety of Spine fusion system manufactured in China is no inferior than imported product.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, comparative, non-inferiority study comparing the change of Japanese Orthopaedic Association Score from baseline at postoperative 24 weeks for patients implanted with local made Spine Fusion System versus imported products.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years old, male or female;
* Subject being diagnosed as having disc degeneration disease, spondylolisthesis, spinal fracture, deformity(degenerative deformity), spinal stenosis, or spinal tumor, has been treated with conservative treatment without relief or getting worse, who is suitable for surgery according to clinic practice.
* Subject is a suitable candidate for implanting investigational products described in study protocols according to investigator's assessment;
* Patient, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and willing to be available for each required study procedure over the study duration.
* Subject has been given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to study Sponsor.

Exclusion Criteria:

* Patient has a local or systemic infection.
* Patient has had one or more previous non-fusion spinal surgery at the involved level(s).
* Patient without spinal deformity and requires fusion at 3 or more levels.
* Has been previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
* Has presence of active malignancy
* Has a medical condition with less than 1 year of life expectancy.
* Pregnancy or women in lactation period.
* Is grossly obese, i.e. Body Mass Index≥40.
* Has a diagnosis, which requires postoperative medication or treatment that interferes with fusion, such as steroids, chemotherapy, radiotherapy, growth factor (for more than 3 months), Nonsteroidal Antiinflammatory Drugs(for more than 3 months), and etc.
* Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g. uncontrolled Diabetes with medication, renal osteodystrophy, or osteogenesis imperfect)
* Alcoholic (taking more than 40g/day, equals to 100ml 50°Chinese liquor), smoking more than 40 cigarettes/day, or Drug abuser;
* Is currently participating in another investigational drug or device study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of Japanese Orthopaedic Association score | Preoperation and 24week post operation
  Questionnaire

SECONDARY OUTCOMES:
Improvement rate of Japanese Orthopaedic Association score | 7day, 12week, and 24week post operation
  Questionnaire
Fixation stability | 12week, and 24week post operation
  Fixation stability should be measured based on translational motion and angular motion which is demonstrated on X-Ray examination (A/P lateral, Flexion and extension).
Visual Analogue Score of low back and leg pain | 7day, 12week, and 24week post operation
  Visual Analogue Scale
Wound healing | 7day, 12week, and 24week post operation
  would healing are classified as 3 classes. (Class I, Class II, Class III)

OTHER OUTCOMES:
Adverse Events | up to 24week post operation
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, Principal Investigator — Beijing Jishuitan Hospital
Locations (8):
- China (8):
  - Anhui Province Hospital, Hefei, Anhui
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University Medical College, Xi’an, Shanxi
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan